CLINICAL TRIAL: NCT06553066
Title: Deep Versus Moderate Neuromuscular Blockade in Bariatric Surgery:
Brief Title: Deep Versus Moderate Neuromuscular Blockade in Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Nikolas Drakos, MD, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bariatric
Record Dates: First submitted 2024-07-04; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: in the assessment of the surgical field quality surgeons are blind respect the level of neuromuscular block received by patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DNMB ( Deep neuromascular blockage) (Experimental): Deep Neuromuscular Block group Intervention: maintenance of a deep neuromuscular block with rocuronium, titrated to maintain a TOF count of 0, and a PTC between 1-2.
  Quality of surgical field conditions' assessed by a blind surgeon as a 5 points scale(Leiden scale : 1 indicates extremely poor conditions, 2 poor conditions, 3 acceptable conditions, 4, good conditions and 5 optimal conditions)
  Interventions: Drug: Deep neuromascular blockage; Drug: Moderate neuromascular blockage
- Group MNMB ( Moderate neuromascular blockage) (Active Comparator): Moderate Neuromuscular Block group Intervention: maintenance of a moderate neuromuscular block with rocuronium, titrated to obtain a TOF count of 1-3.
  Quality of surgical field conditions' assessed by a blind surgeon as a 5 points scale(Leiden scale : 1 indicates extremely poor conditions, 2 poor conditions, 3 acceptable conditions, 4, good conditions and 5 optimal conditions)
  Interventions: Drug: Deep neuromascular blockage; Drug: Moderate neuromascular blockage

INTERVENTIONS:
Drug: Deep neuromascular blockage — maintenance of a deep neuromuscular block with rocuronium, titrated to maintain a TOF count of 0, and a PTC between 1-2.
  Quality of surgical field conditions' assessed by a blind surgeon as a 5 points scale(Leiden scale : 1 indicates extremely poor conditions, 2 poor conditions, 3 acceptable conditions, 4, good conditions and 5 optimal conditions)
  Other Names: Rocuronium and Sugammadex
Drug: Moderate neuromascular blockage — maintenance of a moderate neuromuscular block with rocuronium, titrated to maintain a TOF count of 1-2
  Other Names: Rocuronium and Sugammadex

SUMMARY:
The aim of this study is to investigate the effect of depth of neuromuscular blockade on the surgical field, patient postoperative pain, intestinal motility, the incidence of postoperative nausea and vomiting and the effect of deep versus moderate neuromuscular blockade on postoperative atelectasis quantitatively using chest computed tomography.This is a prospective, randomized, controlled clinical-controlled study in patients ≥18 years old scheduled to undergo elective bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years ASA II-III who are to undergo planned laparoscopic bariatric surgery

Exclusion Criteria:

* ASA 4 patients
* Maternal population
* Patients who are not scheduled to receive general anesthesia, but some other type of anesthesia.
* Contraindicated patients: administration of neuromuscular blockade, suppression of spontaneous respiration, and those with an indication for awake intubation or surgical airway.
* Patients with neuromuscular diseases
* Patients who refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
impact of a deep neuromuscular blockade on surgical conditions | During surgery
  impact of a deep neuromuscular blockade (TOF count = 0 and posttetanic count [PTC] 1-2) and a moderate neuromuscular blockade (TOF count= 1 - 3) on intraoperative surgical conditions assessed by the surgeon as a 5 points scale

SECONDARY OUTCOMES:
the effect of deep versus moderate neuromuscular blockade on postoperative atelectasis quantitatively using chest computed tomography. | in the first six postoperative hours
  quantitatively using chest computed tomography and expressed as percentage to total lung tissue volume
Postoperative pain | first postoperative day
  Pain was measured four times in the PACU (at 15 min intervals starting upon arrival) and twice on the ward (8PM the day of surgery and 2 PM the next day).Pain was measured using an 11-point numerical rating scale (NRS), ranging from 0 (no pain) to 10 (most pain imaginable).
Mean arterial pressure (mmHg) | intraoperative and in Postanesthesia care unit
  measured before induction to general anesthesia, immediately after induction and every 15 min until the end of operation and immediately after awareness.at 15 min intervals starting upon arrival in the post anesthesia care unit
PIPcmH20 ( Peak inspiratory pressure) | intraoperative
  Respiratory mechanical parameters were measured after intubation at suspine position, after insufflation of pneumoperitoneum , then the standard different positions of the patient ( Anti-Trendelenburg, supine, anti-trendelenburg and suspine position without premoperitoneum at the end of the procedure)
duration of surgery (hr) | intrapostoperative
  from the incision to the last skin suture
The first flatus time (min) | up to 5 days
  the first time that patient flatus postoperative
duration of anesthesia time (min) | intraoperative
  time from anesthesia induction to Extubation
Postoperative nausea and vomiting (PONV) | until first postoperative day
  incidence of PONV
Hospitalization time ( days) | up to 2 weeks
  FROM ADMISSION TO HOSPITAL TO DISCHARGE
cumulative analgetid dose (mg) | until 2 PM the next day of the surgery
  cumulative analgetid dose until 2 PM the next day of the surgery
oxygen saturation (SpO2) % | intraoperative and in Postanesthesia care unit
  measured before induction to general anesthesia, immediately after induction and every 15 min until the end of operation and immediately after awareness.at 15 min intervals starting upon arrival in the post anesthesia care unit
tidal volume (ml) | Intraoperative
  Respiratory mechanical parameters were measured after intubation at suspine position, after insufflation of pneumoperitoneum , then the standard different positions of the patient ( Anti-Trendelenburg, supine, anti-trendelenburg and suspine position without premoperitoneum at the end of the procedure)
Pplat cmH20 ( plateau pressure), | Intraoperative
  Respiratory mechanical parameters were measured after intubation at suspine position, after insufflation of pneumoperitoneum , then the standard different positions of the patient ( Anti-Trendelenburg, supine, anti-trendelenburg and suspine position without premoperitoneum at the end of the procedure)
dynamic compliance ml/cmH20, | Intraoperative
  Respiratory mechanical parameters were measured after intubation at suspine position, after insufflation of pneumoperitoneum , then the standard different positions of the patient ( Anti-Trendelenburg, supine, anti-trendelenburg and suspine position without premoperitoneum at the end of the procedure)
DP cmH20( Driving pressure) | Intraoperative
  Respiratory mechanical parameters were measured after intubation at suspine position, after insufflation of pneumoperitoneum , then the standard different positions of the patient ( Anti-Trendelenburg, supine, anti-trendelenburg and suspine position without premoperitoneum at the end of the procedure)
Resistance cmH20/L/sec | Intraoperative
  Respiratory mechanical parameters were measured after intubation at suspine position, after insufflation of pneumoperitoneum , then the standard different positions of the patient ( Anti-Trendelenburg, supine, anti-trendelenburg and suspine position without premoperitoneum at the end of the procedure)
PEEP cmH20 | Intraoperative
  Respiratory mechanical parameters were measured after intubation at suspine position, after insufflation of pneumoperitoneum , then the standard different positions of the patient ( Anti-Trendelenburg, supine, anti-trendelenburg and suspine position without premoperitoneum at the end of the procedure)

IPD SHARING:
Plan to Share IPD: No